CLINICAL TRIAL: NCT06343662
Title: Meraki: Music Therapy Protocol for People with Acquired Brain Injury
Brief Title: Group Music Therapy for Acquired Brain Injury
Acronym: Meraki_ABI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, M. Antonia Pérez-Marín, Associate Professor, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Meraki_Acquired Brain Injury
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Acquired Brain Injury
Keywords: music therapy-based treatment; psychological intervention; discomfort; Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Intervention: Control Group (No Intervention): Patients who receive the treatment program, will previously constitute their own control group (waiting list control group).
- Experimental group (Experimental): Patients admitted to the brain injury unit will participate in a music therapy protocol starting one week after admission. Prior to the group session, three evaluations will be conducted over six days. Post-treatment assessments will also be conducted to enable longitudinal evaluation of the patient over the course of a week.
  Interventions: Behavioral: MERAKI_ABI

INTERVENTIONS:
Behavioral: MERAKI_ABI — The music therapy session will focus on the themes of reidentification and involvement. The aim is to accompany the patient during the illness process, allowing them to express their emotional state, relate to music, promote listening and communication between family members, help and value preserved abilities, and promote personal involvement in the rehabilitation process.
  The session will work with songs, taking into account musical preferences.
  Arms: Experimental group

SUMMARY:
The study aims to analyse the impact of music therapy-based treatment on the comfort and well-being of patients with acquired brain injury (ABI). To achieve this objective, it is proposed to validate and implement a music therapy-based assessment and treatment protocol. The protocol will be tested in a pilot sample to improve adaptation to the disease and promote integration with the usual health measures of patients with ABI. Implementing a group treatment programme based on music therapy applied to patients with ABI.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acquired brain damage who has been admitted to the hospital for at least one week. The patient has experienced a sudden brain injury resulting in physical, psychological, cognitive, behavioural or sensory deficits that have reduced their previous functional capacity and quality of life. The patient is clinically stable enough to undergo rehabilitation and had a good functional situation prior to the episode (Barthel Index > 60).
* Be over 18 years of age.
* The participant or their relatives have signed the informed consent form.
* They have completed the group music therapy intervention session, as well as the pre-test and post-test evaluations.

Exclusion Criteria:

* Failure to obtain informed consent
* The Barthel Index score is below 60, indicating functional dependency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in Discomfort ( Baseline (3 Assessments), Pre- Post) | Baseline up to 1 week
  The Discomfort Observation Scale (DOS) is a tool used to assess discomfort in patients with severe cognitive impairment in end-of-life situations. The Discomfort Observation Scale (DOS) is a tool used to assess discomfort in patients with severe cognitive impairment in end-of-life situations. The Discomfort Observation Scale (DOS) is a tool used to assess discomfort in patients with severe cognitive impairment in end-of-life situations. It consists of nine items that evaluate factors such as noisy breathing, body language, facial expressions, and verbalizations. Each observation is scored dichotomously (0-1, presence-absence), resulting in a score range of 0 to 9. A higher score indicates less discomfort. The language used is clear, concise, and objective, adhering to formal register and precise word choice. The text is grammatically correct and follows conventional structure and formatting features.

SECONDARY OUTCOMES:
Barthel Index | Baseline
  The purpose of this assessment is to evaluate the patient's functional independence. It involves assessing their ability to perform 10 activities of daily living, including eating, washing, dressing, grooming, bowel movements, urination, toileting, transferring, ambulation, and stair use. The scores range from 0, indicating maximum dependence, to 100, indicating maximum independence.
Pfeiffer Short Form Mental State Questionnaire, SPMSQ | Baseline
  This assessment evaluates cognitive impairment through a series of 10 questions that explore orientation, remote and working memory, as well as calculation skills. Each incorrectly answered question adds one point, and more than 2 errors suggest the presence of cognitive impairment that requires further study.
Charlson Comorbidity Index (CCI), | Baseline
  This tool predicts the one-year mortality rate for patients with various comorbid conditions, including heart disease, AIDS, and cancer (a total of 8 conditions in the short version). The measure assigns a score to each condition based on the associated risk of death. A score of 0 to 1 indicates no comorbidity, 2 points indicates low comorbidity, and 3 points or more indicates high comorbidity. The total score predicts mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Marián Pérez-Marín, PhD, Principal Investigator — University of Valencia
Locations (1):
- Hospital Dr. Moliner, Serra, Valencia, Spain